CLINICAL TRIAL: NCT06742619
Title: OBESE PATIENTS AND ANAESTHESİA İNDUCTİON: PERFUSION INDEX, PRONE ,SUPİNE AND SITTING POSITION
Brief Title: PERFUSION INDEX, PRONE ,SUPİNE AND SITTING POSITION
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Other Study IDs: u1103
Record Dates: First submitted 2024-11-18; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Perfusion Index
Keywords: perfusion index; prone; supine; anesthesia
MeSH Terms: conditions — Deception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- gruops: patient supine position
- groupp: patient prone position
- grupsitting: patient sitting position

SUMMARY:
The aim was to investigate the effect of anesthesia management on perfusion index changes in obese patients and different anesthesia positions. The effect of positional intra-abdominal pressure and lung-related variables was investigated.

DETAILED DESCRIPTION:
There may be changes in haemodynamic findings in patients after anaesthesia. The most common of these are hypotension and bradycardia. Many factors play a role on the hypotensive effect of anaesthesia induction1 . Position changes in patients during surgery in obese patients affect these changes.In our study, the changes in haemodimaic findings and the changes in PI and PVI were investigated in patients with BMI 30 and above and in patients with BMI within normal limits after induction of anaesthesia by giving prone position and sitting position.Position changes in patients during surgery in obese patients affect these changes. Hypertension and hypotension after induction of anaesthesia are common in obese patients. In addition, decreased venous return to the heart due to increased intrathoracic pressure during mechanical ventilation may trigger bradycardia and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years range
* Patients who will be operated in supine prone and sitting positions

Exclusion Criteria:

* Heart Failure
* antiarrhythmic drug use hemodynamic instability uncooperative patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be operated in supine prone and sitting positions
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Group P-S-ST | preoperative 5 minute and after anesthesia induction 10 20 30. mimute Perfusion İndex value)
  Comparison after anesthesia induction in prone, supine and sitting positions.(Perfusion index value)

SECONDARY OUTCOMES:
Body mass index, age,comorbidities | preoperative perion (10 minutes before anesthesia)
  in preoperative period patiens body mass index (kg/m2), age (years) and comorbidities were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Hospital, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Many studies can be done due to sharing

REFERENCES:
- [Result] Hara K, Ichihara K, Yamaguchi M, Takeshita H, Kuroki T. Effect of intraoperative operating table rotation on lower limb perfusion index in patients in the lithotomy position. Medicine (Baltimore). 2022 Sep 23;101(38):e30412. doi: 10.1097/MD.0000000000030677. PMID 36197219